CLINICAL TRIAL: NCT04906278
Title: Sequential Use of Foley Catheter With Amniotomy for Second-trimester Pregnancy Termination
Brief Title: Amniotomy for Second-trimester Pregnancy Termination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AM-FO
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Abortion, Missed
MeSH Terms: conditions — Abortion, Missed | interventions — Amniotomy; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amniotomy group (Other): Amniotomy will be performed by toothed forceps. The handle of the device will be held with one hand outside the vagina while 2 fingers of the opposite hand will be placed in the vagina to guide the tip.
  Interventions: Device: Foley catheter balloon; Procedure: Amniotomy; Drug: Oxytocin
- No-amniotomy group (Other): No-amniotomy will be done
  Interventions: Device: Foley catheter balloon; Drug: Oxytocin

INTERVENTIONS:
Device: Foley catheter balloon — A Cusco speculum will be placed and a 16F Foley catheter will be inserted into the cervix using ring forceps. Then the balloon will be inflated with 40 ml of saline and it will be pulled out to ensure the balloon covered the internal os of the cervix
Procedure: Amniotomy — Amniotomy will be performed by toothed forceps. The handle of the device will be held with one hand outside the vagina while 2 fingers of the opposite hand will be placed in the vagina to guide the tip. Care should be taken to protect maternal vaginal tissues from the forceps. Once the forceps reach the amniotic sac, the tip is pushed up against the sac with the index or middle finger of the internal hand to pierce the membranes. The nature of amniotic fluid will be checked.
  Arms: Amniotomy group
Drug: Oxytocin — The intravenous oxytocin infusion will be administered as 10 IU oxytocin/ 500 ml glucose/ 30 mIU/minute were every 6 hours till complete abortion occurs.

SUMMARY:
The termination of abortion is an important issue that has many controversies. The most common time of serious abortion-related complications is the second trimester. Missed abortion is one of the most common indications of termination of pregnancy in the second trimester. Misoprostol and mifepristone are effective drugs for induction of abortion but these drugs are now expensive, and non-available in many developing countries.

The effectiveness of Foley's catheter balloon on cervical ripping for mid-trimester pregnancy termination has been proved before. It can effectually shorten the time of the expulsion of the fetus. Amniotomy defines as an artificial rupture of the membranes; it is an ordinary obstetric practice used mainly in the induction of labor, with good results and less morbidity. The obstetricians used to combine amniotomy with other methods such as prostaglandins or oxytocin to induce labor in a woman with an unfavorable cervix.

Despite plenty of studies that investigated the role of amniotomy for induction of labor but the studies which addressed the role of amniotomy in the induction of second-trimester abortion are very scarce in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40 years old.
* Women who are pregnant in singleton mid-trimester missed abortion (18-26 weeks).
* Bishop's score is ≤ 4.

Exclusion Criteria:

* Women who delivered before by classic caesarian section or had a history of -myomectomy, hysteroscopic uterine surgery, or cervical surgery like conization.
* Women with multiple gestations.
* Women with ultrasonography evidence of low amniotic fluid volume.
* Women with rupture of fetal membranes.
* Women with evidence of low implanted placenta by ultrasound.
* History or laboratory evidence of intra-uterine infection.
* History is suggestive of latex allergy.
* Women with severe anemia, hypertension, diabetes, or with coagulopathy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
The interval between induction to complete abortion | 15 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided